CLINICAL TRIAL: NCT05881902
Title: THE EFFECT OF CANCER EDUCATION BASED ON THE HEALTH BELIEF MODEL ON AWARENESS OF WOMEN WITH DISABILITIES AND THEIR PARTICIPATION IN SCREENING
Brief Title: THE EFFECT OF CANCER EDUCATION ON WOMEN'S AWARENESS LEVELS AND THEIR BEHAVIORS ON SCREENINGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeşim KAYAPA (Other)
Responsible Party: Sponsor-Investigator, Yeşim KAYAPA, PhD student, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: AYBÜ-HMS-YK-01
Record Dates: First submitted 2023-02-27; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Cancer
Keywords: cancer screening; cancer early detection; physically disabled; early screening; health blief model; breast cancer; cervix cancer; awareness
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant, Outcomes Assessor
Masking Description: The collected data will be analyzed by an independent statistician. The fact that the intervention 1 and intervention 2 groups of the study are known by the researcher and the women with physical disabilities do not know, makes it a double-blind randomized controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention 1: Cancer awareness training based on the Health Belief Model (Experimental): Awareness training based on the Health Belief Model will be given to the participants in the Intervention 1 group during home visits in order to eliminate the lack of information about the common female cancers in women and to increase their awareness. For 3 months, intervention 1 group will be given applications to reinforce their awareness in the education based on the Health Belief Model (for BSE and KKVM, erasable calendar magnets, booklets, phone cases and accessories themed as "common cancers awareness in women" as a reminder, phone call) will be made.
  Interventions: Behavioral: HEALTH FAITH MODEL GUIDED IN CANCER FREQUENTLY SEEN IN WOMEN EARLY DIAGNOSIS AND SCREENING METHODS EDUCATION
- İntervention 2: Standart cancer education (Experimental): Participants in the Intervention 2 group will be provided with the standard training applied at KETEM by the Ministry of Health on female cancers, which are frequently seen in physical women, during home visits. The training will be held in the form of power-point presentation, question and answer. For 3 months, intervention 2 groups will be applied to reinforce their awareness in standard education (sms reminder).
  Interventions: Behavioral: STANDART CANCER EDUCATİON

INTERVENTIONS:
Behavioral: HEALTH FAITH MODEL GUIDED IN CANCER FREQUENTLY SEEN IN WOMEN EARLY DIAGNOSIS AND SCREENING METHODS EDUCATION — A total of 4 home visits and 2 phone calls will be made by giving awareness training based on the Health Belief Model to the participants in the Intervention 1 group in order to eliminate the lack of information about the common female cancers in women and to increase their awareness. For 3 months, intervention 1 group will be given applications to reinforce their awareness in the education based on the Health Belief Model (for BSE and KKVM, erasable calendar magnets, booklets, phone cases and accessories themed as "common cancers awareness in women" as a reminder, phone call) will be made
  Arms: İntervention 1: Cancer awareness training based on the Health Belief Model
Behavioral: STANDART CANCER EDUCATİON — The participants in the intervention 2 group will be given the standard training applied by the Ministry of Health in KETEM for women's cancers during home visits, and a total of 4 home visits and 2 SMS reminders will be made.
  Arms: İntervention 2: Standart cancer education

SUMMARY:
Disability is part of being human. He estimates that the prevalence of disability among women is 60% higher than that of men.

Disabled women coexist in a dual state of vulnerability where "being a woman" and "being a disabled person" have two social disadvantages. Among people with disabilities, women with disabilities (WWD) have higher unmet healthcare needs than women without disabilities.

Cancer is an important public health problem and cause of death all over the world. Among the most common cancers in women; breast, uterine corpus, ovarian and cervix cancers are seen to be prominent, respectively. It is known that with regular examinations and screenings, early diagnosis of breast and cervical cancer increases the chance of treatment.

International studies show that women face barriers and difficulties in accessing reproductive health and cancer screening services. In studies, it was stated that especially women with disabilities living in rural areas had lower mammography and Pap-smear tests compared to women without disabilities. In recent years, the Health Belief Model has been used frequently to examine the effect of health beliefs on cancer screening behaviors in women and to increase screening rates. The model explains the beliefs and attitudes that affect individuals' behaviors. According to the model; If a person has a desire to prevent illness or a belief in recovery, he recommends taking a specific health action to prevent illness as a positive behavior. It was emphasized that nurses have important roles and responsibilities in the protection and development of health, and that they can identify individuals with disabilities who are considered "fragile", and provide health education and counseling to these groups. It is thought that the "disabled-friendly accessible health care" practices under the guidance of the Health Belief Model will bring the preventive health care behavior of women with disabilities to the desired level.

Disabled women experience inequalities in benefiting from routine health services and health screening services in special areas such as reproductive health and protection from women's cancers. Being diagnosed with cancer is undoubtedly devastating for anyone. For this reason, it becomes more important to raise awareness about the prevention, prevention, early diagnosis and development of a healthy lifestyle in women with physical disabilities, and to encourage health-seeking behaviors.

DETAILED DESCRIPTION:
Disability is part of being human. Everyone may be temporarily or permanently disabled at some point in their life, and it has been stated that they will experience increasing difficulties in functioning in old age. He estimates that the prevalence of disability among women is 60% higher than that of men.

Disabled women coexist in a dual state of vulnerability where "being a woman" and "being a disabled person" have two social disadvantages. Among people with disabilities, women with physical disabilities have higher unmet healthcare needs than women without disabilities.

Cancer is an important public health problem and cause of death all over the world. According to the Turkish Cancer Statistics, it is estimated that approximately 69,633 women are diagnosed with cancer in our country. Among the most common cancers in women; breast, uterine corpus, ovarian and cervix cancers are seen to be prominent, respectively. It is known that with regular examinations and screenings, early diagnosis of breast and cervical cancer increases the chance of treatment.

International studies show that women face barriers and difficulties in accessing reproductive health and cancer screening services. In the study of Horner-Johson et al., it was stated that especially rural women with disabilities had lower mammography and Pap-smear tests compared to non-disabled women. It is emphasized that as a result of lower screening participation of persons with disabilities, there is a higher risk of cancer mortality with delayed diagnosis.

In another study investigating the reasons why women with physical disabilities do not engage in preventive health services; time constraints and priorities, interactions between health professionals and women with disabilities, lack of knowledge, belief, sensitivity, belief that people with disabilities have more information than service providers, economic problems, transportation problems, appointment problems, availability of accessible facilities, physical pain, mammography, pap smear It has been stated that factors such as both psychological and physical discomfort during the test and pelvic examination are effective.

In recent years, the Health Belief Model (SIM) has been frequently used to examine the effect of health beliefs on cancer screening behaviors in women and to increase screening rates. The model explains the beliefs and attitudes that affect the behavior of individuals. The most basic components of the model are the perception of susceptibility, the perception of seriousness, the perception of benefit, the perception of obstacles, the health motivation and the perception of trust. The SIM recommends that if a person has a desire to prevent illness or a belief in recovery, he or she should take a specific health action to prevent illness as a positive behavior. In an interventional study conducted with Korean-American women to improve breast cancer screening, using SIM for early diagnosis and behavioral change, it was determined that the rate of mammography and Breast Self-Examination (BSE) application rates increased significantly. It has been emphasized that nurses have important roles and responsibilities in the protection and development of health, and that they can identify disabled individuals who are considered "fragile" and provide health education and counseling to these groups. It is thought that awareness training on cancers that are common in women, given under the guidance of the Health Belief Model, will bring the preventive health behavior of women with disabilities to the desired level. When the literature is examined, the limited number of randomized controlled studies that will increase the participation of disabled women in cancer screening services increases the importance of the subject.

Disabled women experience inequalities in benefiting from routine health services and health screening services in special areas such as reproductive health and protection from cancers that are common in women. Being diagnosed with cancer is undoubtedly devastating for anyone. For this reason, it becomes more important to raise awareness about the prevention, prevention and early diagnosis of cancers that are common in women with physical disabilities, to raise awareness on this issue and to encourage health-seeking behaviors.

This study was conducted to determine the barriers for women with physical disabilities between the ages of 18-65 to adopt behaviors to diagnose common cancers in women at an early stage, and to increase participation in early diagnosis behaviors in cancers that are common in women (Breast Self Examination (BSE), Clinical Breast Examination (CBE), Self-Examination). Vulva Self Examination (KKVM), Mammography and PapSmear Test) was planned to determine the effectiveness of awareness training based on SIM.

ELIGIBILITY:
Inclusion Criteria:

* Being physically disabled
* Having a disability to perform KKMM and KKVM
* Being between the ages of 18-65 (since these are the age ranges at which screening is started),
* Being married or living with a spouse (for participation in cervical cancer screening),
* Not to do KKMM and KKVM regularly every month,
* Never or in the last three years have not had a pap smear test, CMM or mammography,
* Not being pregnant, breastfeeding or postpartum,
* Not having a history of common cancers in women,
* Accepting to participate in the research,
* Being literate, accessible and communicative,
* Absence of severe psychiatric problems

Exclusion Criteria:

* Hearing impairment
* Being visually impaired
* Being mentally handicapped
* A physically disabled woman who gives up working at any stage of the study will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Our sample is considered based on biological sex.
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The Gynecological Cancers Awareness Scale | 12 weeks
  The Gynecological Cancers Awareness Scale consists of 41 questions in total, with a minimum of 41 and a maximum of 205 points that can be obtained from the scale. The increase in the scores obtained from the scale indicates that the awareness of gynecological cancer increases.

SECONDARY OUTCOMES:
Champion's Health Belief Model Scale for Breast Cancer and Screening | 12 weeks
  In the scale, 2 sub-dimensions will be used that question the "barriers" of performing breast self-examination and the "barriers" of mammography. Higher scores indicate that obstacles are perceived as high for the perception of obstacles.

OTHER OUTCOMES:
Cervical Cancer and Pap-Smear Test Health Belief Model Scale | 12 weeks
  women with cervical cancer and perceptions of their health beliefs about the Pap Smear test. (their susceptibility to cervical cancer, perceptions of its severity, Pap smear about the benefits of having a test or the barriers to getting this test done. perception) measures the effect of having Pap smears.
Evaluation Form for Participation in Screening of Common Cancers in Women | 12 weeks
  The form determines the rates of women performing breast self-examination, clinical breast examination, mammography, self-vulva examination and pap-smear during the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be used in metaanalysis research, but provided that you receive an information mail.